CLINICAL TRIAL: NCT07124325
Title: The Use of Remote Cardiotocography Telemonitoring Within High-risk Pregnancy Care.
Brief Title: Remote Cardiotocography Telemonitoring Within High-risk Pregnancy Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Jack Hamer, Clinical research fellow, Birmingham Women's NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 27-6-194
Record Dates: First submitted 2025-08-01; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy; High Risk; Telemonitoring; Telemedicine; Cardiotocography

STUDY DESIGN:
Intervention Model Description: 50 participants split in one arm using the home CTG device. To detect a 20% difference in the mean anxiety scores pre- and post-study a sample size with a power of 90% (α =0.05), a sample size of 42 is required. 50 recruited women will allow for a 10% drop out rate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home antenatal CTG monitoring (Experimental): Participants will be asked to use the remote monitoring devices one a week for a 1 hour each time for up to 6 weeks or until delivery.
  Participants are eligible if they are aged 18 over over, 32+0 gestation onwards, singleton pregnancy, able to speak English and have at least one of 6 high-risk pregnancy conditions.
  Interventions: Device: Pregnabit Pro device and PregnaOne platform

INTERVENTIONS:
Device: Pregnabit Pro device and PregnaOne platform — Remote CTG device and online dashboard for remote pregnancy care

SUMMARY:
The overall aim of this research proposal is to explore the feasibility and acceptability of home antenatal maternal-fetal monitoring technology within a high-risk pregnancy group. The investigators hypothesise that home monitoring is feasible and acceptable to both pregnant women and HCPs.

50 women from a single site will be recruited to use a home cardiotocography (CTG) device alongside routine antenatal care. Participants will use this device once a week, for an hour at a time, for up to 6 weeks or until delivery. The primary outcome is 20 minutes of continuous monitoring. Additional outcomes assess acceptability, adherence and safety.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 years
* Gestational age 32+0 weeks onwards.
* Singleton pregnancy.
* Able to speak English
* Receiving antenatal care which includes routine antenatal fetal monitoring for one of the 6 index conditions (hypertensive disease in pregnancy, reduced fetal growth (small for gestational age and fetal growth restriction) obstetric cholestasis, PPROM, previous history of stillbirth and recurrent reduced fetal movements )
* Able to give written informed consent.
* Willing to attend hospital immediately in the event of an unexpected finding whilst using the home devices.

Exclusion Criteria:

* Multiple pregnancy.
* Fetal abnormalities or a non-viable fetus.
* Body mass index (BMI) ≥35
* Women with internal cardiac devices such as pacemaker and implantable cardioverter defibrillator.
* History of allergic reaction to skin adhesives and/or latex.
* Acute or chronic skin lesions and wounds in areas in contact with the device.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The number of participants that produce interpretable antenatal maternal-fetal monitoring cardiotocogram (CTG) traces for each episode of intermittent home monitoring. | Through study completion, an average of 9 months
  Completion of an at least 20 minutes of uninterrupted interpretable fetal heart recording which has computerised capability. This will be defined as a percentage derived from the number of monitoring episodes achieving the primary outcome divided by the total number of monitoring episodes.

SECONDARY OUTCOMES:
The number of participants completing the full schedule of home maternal-fetal monitoring episodes. | Through study completion, an average of 9 months
  Determined as the median number of monitoring episodes completed.
The number of women approached who agreed to participate within the study. | Pre-intervention
  Number participants agreeing out of total women approached
What are the emotions of participants using home maternal-fetal monitoring. | Pre-intervention
  Pre-intervention questionnaire using the accredited STAI anxiety questionnaire.
What are the emotions of participants using home maternal-fetal monitoring and is there an impact before and after a singular monitoring episode? | Through study completion, an average of 9 months
  Questionnaire using the accredited STAI anxiety questionnaire at several time points whilst using the home monitoring device. Results compared pre and post monitoring episode to determine a if there is a discriminative impact on anxiety scores whilst using the home monitoring device. Results will be displayed graphically and compared using P value.
What are the emotions of participants using home maternal-fetal monitoring and was there any change from the beginning of the study. | Immediately after the intervention
  Post-intervention questionnaire using the accredited STAI anxiety questionnaire. Results compared to the scores at the beginning of the study and demonstrated graphically and with a P value.
The usability of the remote monitoring device. | Immediately after the end of the intervention
  Assessed post study using the validated system usability scale scoring questionnaire.
The number of participants with unexpected clinical outcomes detected whilst using home monitoring devices, which warrants patients to attend maternity triage for assessment and/or modification of ones antenatal care. | Through study completion, an average of 9 months
  Number of unexpected outcomes requiring attendance to triage out of total number of monitoring episodes, presented as a percentage.
What are the views of participants regarding acceptability of home maternal-fetal monitoring. | Pre-intervention
  Pre-intervention questionnaire using a 5 point Likert Scale (range from Strongly agree on the left, to strongly disagree on the right). No total score, each question individual and a tick box.
What are the views of participants regarding acceptability of home maternal-fetal monitoring. | Immediately after the intervention
  Post-intervention questionnaire using a 5 point Likert Scale (range from Strongly agree on the left, to strongly disagree on the right). No total score, each question individual and a tick box.
The influence of participant demographics on achieving the primary outcome. | Through study completion, an average of 9 months
  Analysis of factors which may influence achievement of the primary outcome. This includes ethnicity, education level, fetal presentation, parity. Presented as event numbers to calculated odds ratio's.
Determining participant adherence to commencing the monitoring episodes | Through study completion, an average of 9 months
  Defined as the median time between when the participant commencing the monitoring episode and the time originally agreed to commence the monitoring episode previously jointly agreed between the researchers and participant.
The influence of fetal movements on achieving the primary outcome | Through study completion, an average of 9 months
  Analysis of fetal movements during a monitoring episode and its influence on the primary outcome. Number of movements in the group achieving primary outcome compared to the group not achieving the primary outcome will be compared using the student T test.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Hamer, MBChB, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust
Locations (1):
- Birmingham Women's and Children's NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No